CLINICAL TRIAL: NCT07382245
Title: Efficacy of Silver Diamine Fluoride Versus Nano-Silver Fluoride in Arresting Active Dentin Caries in Primary Teeth in Young Children: A Randomized Clinical Trial
Brief Title: Efficacy of Silver Diamine Fluoride Versus Nano-Silver Fluoride in Arresting Active Dentin Caries in Primary Teeth in Young Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: October University for Modern Sciences and Arts (Other)
Responsible Party: Principal Investigator, khaled sayed, lecturer assistant at pediatric dentistry department- faculty of dentistry- October University for Modern Sciences and Arts -, October University for Modern Sciences and Arts
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Khaled SDF
Record Dates: First submitted 2026-01-25; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Early Childhood Caries (ECC); Active Dentin Caries in Primary Molars
Keywords: Early Childhood Caries; primary molar; Nano-Silver Fluoride; Silver Diamine Fluoride; SDF
MeSH Terms: interventions — silver diamine fluoride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Nano-Silver Fluoride (Experimental): Topical application of Nano-Silver Fluoride varnish containing silver nanoparticles, chitosan, and fluoride applied to active dentin caries lesions in primary molars. Application will be performed twice: at baseline and after 6 months, without caries excavation or restoration.
  Interventions: Drug: Nano-Silver Fluoride
- Arm B: Silver Diamine Fluoride (Active Comparator): Topical application of 38% Silver Diamine Fluoride varnish applied to active dentin caries lesions in primary molars. Application will be performed twice: at baseline and after 6 months, without caries excavation or restoration.
  Interventions: Drug: Silver Diamine Fluoride

INTERVENTIONS:
Drug: Nano-Silver Fluoride — Chitosan (28,585 μg/ml), Silver (376.5 μg/ml) and Sodium fluoride (5028.3 μg/ml)
  Arms: Arm A: Nano-Silver Fluoride
Drug: Silver Diamine Fluoride — 38% Silver Diamine Fluoride
  Arms: Arm B: Silver Diamine Fluoride

SUMMARY:
Early childhood caries is a major public health problem affecting preschool children worldwide. Silver Diamine Fluoride is a well-established non-invasive treatment for arresting caries; however, it causes black discoloration of treated lesions. Nano-Silver Fluoride has been introduced as an alternative that may arrest caries without discoloration.

This randomized clinical trial aims to compare the efficacy of Silver Diamine Fluoride and Nano-Silver Fluoride in arresting active dentin caries in primary teeth and to assess discoloration, post-operative pain, and parental satisfaction over a 12-month follow-up period.

DETAILED DESCRIPTION:
This randomized clinical trial will be conducted on 30 children aged 3-5 years attending the outpatient clinic of Pediatric Dentistry, Faculty of Dentistry, Suez Canal University. Children with active dentin caries in primary molars will be randomly allocated into two groups: Silver Diamine Fluoride group and Nano-Silver Fluoride group.

Both materials will be applied topically without caries excavation. Clinical evaluation will be performed at baseline and at 1, 3, 6, 9, and 12 months using ICDAS criteria, visual and tactile examination, assessment of post-operative pain, discoloration through standardized photographs, and parental satisfaction questionnaires.

The primary outcome is caries arrest. Secondary outcomes include discoloration, pain, and parental satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy children.
* Children with age ranged from 3-5 years from both genders.
* Children who refused dental treatment with Frankl Behavior Rating Scale 1 and 2.
* Children having molars with active dentin caries score (2,3,4) according to International Caries Detection and Assessment System- ICDAS II, detected by visual and tactile.
* Parents/guardians accept treatment and write informed consent.

Exclusion Criteria:

* Children with allergy to silver from their medical history.
* Children with ulcerative gingivitis.
* Children with primary molars with the following criteria:
* Symptomatic
* Involving the pulp
* Presence of fistula or sinus
* Presence of gingival inflammation and Pain on percussion
* Close to exfoliation

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-02-25 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Caries arrest of active dentin caries | 1, 3, 6, 9 and 12 months
  Arrest of caries assessed clinically by hardness of dentin using blunt periodontal probe and ICDAS criteria

SECONDARY OUTCOMES:
Discoloration of carious lesions | 1, 3, 6, 9 and 12 months
  Assessment of color change using standardized pre- and post-operative photographs
Post-operative pain | 1, 3, 6, 9 and 12 months
  Presence or absence of pain assessed through parental interview
Parental satisfaction | 1, 3, 6, 9 and 12 months
  Evaluation using a structured parental satisfaction questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, MSA University, Giza, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes